CLINICAL TRIAL: NCT02246829
Title: Assessment of Early Changes in SD-OCT After Initiation of a Treatment by Intravitreal Aflibercept (EYLEA®) (2mg) Over a 12-week Period for Patients Suffering From Neovascular Age-related Macular Degeneration (AMD) French SD OCT in wAMD
Brief Title: Assessment of Early Changes in SD-OCT After Initiation of a Treatment by Intravitreal Aflibercept (EYLEA®)START
Acronym: START
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2013/18
Record Dates: First submitted 2014-09-11; First posted 2014-09-23 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Neovascular Age-related Macular Degeneration of All Subtypes
Keywords: wet AMD, SD-OCT, intravitreal injection, central retinal thickness,
MeSH Terms: interventions — Intravitreal Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept 2mg Intravitreal injection (Other): 2 mg intravitreal Aflibercept initiated with one injection every 4 weeks for three consecutive doses (loading dose) The duration of the follow-up is 12 weeks. This means 3 injections per patient should be given over the study period
  Interventions: Procedure: Intravitreal injection

INTERVENTIONS:
Procedure: Intravitreal injection — 2 mg intravitreal Aflibercept initiated with one injection every 4 weeks for three consecutive doses (loading dose) The duration of the follow-up is 12 weeks. This means 3 injections per patient should be given over the study period

SUMMARY:
Aflibercept (EYLEA®) induces a rapid reduction in central retinal thickness (CRT) for patients suffering from neovascular age-related-macular degeneration.1 This early dramatic reduction in CRT is already observed through week 4. Therefore it might be not necessary to consistently perform each of the three monthly consecutive intravitreal injections of the so-called loading phase.

DETAILED DESCRIPTION:
The aim of this study is to assess whether the retina of some patients has dried up after the first or second intravitreal injection of Aflibercept (EYLEA®) 2mg and in that event, to determine the proportion of these patients The analysis of the characteristics could help identify a morphotype that would predict whether and when the retina will dry up within the first 3 months of treatment. For some patients having an early drying-up, the third monthly injection might be not necessary 50 naïve patients will be included and will receive a monthly injection over 12 weeks with a biweekly follow-up. Morphological and functional characteristics will be recorded at each visit and will be analyzed. The rate of patients with dry SD-OCT will be assessed.

The study includes 7 visits. The visits are scheduled on an every 2-week basis from baseline to Week 12. V1 (baseline), V3 and V5, the patient will be injected with Aflibercept (EYLEA®) 2mg. In the other visits, the visual acuity test, Fundus photography, SD-OCT, and/or Fluorescein Angiography are performed

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 50 years of age
* Active primary subfoveal choroidal neovascularization (CNV) lesions secondary to AMD including juxtafoveal lesions that affects the fovea as evidenced by FA in the study eye
* Signed Informed Consent
* Willing, committed, and able to return for ALL clinic visits and complete all study-related procedures.

Exclusion Criteria:

* Prior treatment with anti-VEGF therapy in the study eye
* Active or suspected ocular or periocular infection.
* Active severe intraocular inflammation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Occurence of a Dry SD-OCT 12-week after initiation of a treatment by Aflibercept (EYLEA®) 2mg | 12-week after initiation of a treatment by Aflibercept (EYLEA®) 2mg

SECONDARY OUTCOMES:
Time to get a dry SD-OCT after initiation of a treatment by Aflibercept | Every 2 weeks from treatment initiation (inclusion) to week 12
Evolution of morphological and visual modification under Aflibercept (EYLEA®) | Every 2 weeks from treatment initiation (inclusion) to week 12
Occurence of pigment epithelial detachment | Every 2 weeks from treatment initiation (inclusion) to week 12
Evolution of retinal hemorrhage if any | Every 2 weeks from treatment initiation (inclusion) to week 12
Evolution in the atrophic lesions | Every 2 weeks from treatment initiation (inclusion) to week 12
Occurence the central Retinal Thickness | Every 2 weeks from treatment initiation (inclusion) to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François KOROBELNIK, Professor, Principal Investigator — University Hospital Bordeaux, France; Geneviève CHENE, MDPhD, Study Chair — University Hospital Bordeaux, France
Locations (10):
- France (10):
  - Service d'ophtalmologie Hôpital Henri Mondor 40, avenue de Verdun, Créteil
  - Service Ophtalmologie CHU DIJON 14 rue Gaffarel BP 77908, Dijon
  - Service d'Ophtalmologie Hôpital de la croix rousse, Lyon
  - Cabinet d'ophtalmologie 1 rue Pougin de la Maisonneuve, Montargis
  - Sce Ophtalmologie CHU Nantes 1 place Alexis Ricordeau, Nantes
  - Centre ophtalmique d'imagerie et de laser (CIL) 11 rue Antoine Bourdelle, Paris
  - Sce du Pr SAHEL Fondation ROTHSCHILD 25 rue Manin, Paris
  - Sce Ophtalmologie Hôpital Lariboisière 2 rue Ambroise Paré, Paris
  - Service Opthalmo 2 Clinique Mathilde 4 rue de Lessard, Rouen
  - Centre Ophtalmologie Transparence 30 Boulevard Heurteloup, Tours

REFERENCES:
- [Background] Patel KH, Chow CC, Rathod R, Mieler WF, Lim JI, Ulanski LJ 2nd, Leiderman YI, Arun V, Chau FY. Rapid response of retinal pigment epithelial detachments to intravitreal aflibercept in neovascular age-related macular degeneration refractory to bevacizumab and ranibizumab. Eye (Lond). 2013 May;27(5):663-7; quiz 668. doi: 10.1038/eye.2013.31. Epub 2013 Apr 5. PMID 23558214
- [Background] Cruess AF, Zlateva G, Xu X, Soubrane G, Pauleikhoff D, Lotery A, Mones J, Buggage R, Schaefer C, Knight T, Goss TF. Economic burden of bilateral neovascular age-related macular degeneration: multi-country observational study. Pharmacoeconomics. 2008;26(1):57-73. doi: 10.2165/00019053-200826010-00006. PMID 18088159
- [Background] Rosenfeld PJ, Brown DM, Heier JS, Boyer DS, Kaiser PK, Chung CY, Kim RY; MARINA Study Group. Ranibizumab for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1419-31. doi: 10.1056/NEJMoa054481. PMID 17021318
- [Background] Cohen SY, Souied EH, Weber M, Dupeyron G, de Pouvourville G, Lievre M, Ponthieux A. Patient characteristics and treatment of neovascular age-related macular degeneration in France: the LUEUR1 observational study. Graefes Arch Clin Exp Ophthalmol. 2011 Apr;249(4):521-7. doi: 10.1007/s00417-010-1553-0. Epub 2010 Nov 6. PMID 21057805
- [Background] Heier JS, Boyer D, Nguyen QD, Marcus D, Roth DB, Yancopoulos G, Stahl N, Ingerman A, Vitti R, Berliner AJ, Yang K, Brown DM; CLEAR-IT 2 Investigators. The 1-year results of CLEAR-IT 2, a phase 2 study of vascular endothelial growth factor trap-eye dosed as-needed after 12-week fixed dosing. Ophthalmology. 2011 Jun;118(6):1098-106. doi: 10.1016/j.ophtha.2011.03.020. PMID 21640258
- [Derived] Korobelnik JF, Souied EH, Oubraham H, Razavi S, Mauget-Faysse M, Savel H, Chene G, Wolf S. ASSESSMENT OF EARLY CHANGES IN SPECTRAL DOMAIN-OPTICAL COHERENCE TOMOGRAPHY AFTER INITIATION OF TREATMENT WITH INTRAVITREAL AFLIBERCEPT (EYLEA) OVER A 12-WEEK PERIOD FOR PATIENTS WITH NEOVASCULAR AGE-RELATED MACULAR DEGENERATION: A Multicenter French Study (START). Retina. 2021 Mar 1;41(3):588-594. doi: 10.1097/IAE.0000000000002910. PMID 33600134